CLINICAL TRIAL: NCT03640351
Title: Clinical Effects of Diquas-S for Patients With Dry Eye After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0601
Record Dates: First submitted 2018-07-23; First posted 2018-08-21 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Dry Eye; Cataract Surgery
Keywords: Dry eye; Cataract surgery; Diquas; preservative free
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Methods: The subjects are randomly divided into three groups. Group 1 uses preservative diquafosol ophthalmic solution, Group 2 uses preservative containing diquafosol ophthalmic solution, and Group 3 uses preservative free sodium hyaluronate after cataract surgery. Before surgery, all patients underwent a detailed ophthalmological examination that included slit-lamp examination (Haag-Streit, Köniz, Switzerland), and dry eye parameters including tear breakup time (TBUT), schirmer test, ocular surface disease index (OSDI), and MGD staging. Corneal wavefront aberrations were measured using i-Trace (Tracey Technologies Corp. Houston, TX). All examinations were repeated at 1, and 3 months after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preservative free diquafosol group (Active Comparator): The subjects use preservative free diquafosol ophthalmic solution after cataract surgery
  Interventions: Drug: 1. Use of preservative free diquafosol ophthalmic solution after cataract surgery
- Preservative containing diquafosol group (Active Comparator): The subjects use preservative containing diquafosol ophthalmic solution after cataract surgery
  Interventions: Drug: 2. Use of preservative containing diquafosol ophthalmic solution after cataract surgery
- Preservative free sodium hyaluronate group (Active Comparator): The subjects use preservative free sodium hyaluronate ophthalmic solution after cataract surgery
  Interventions: Drug: 3. Use of preservative free sodium hyaluronate ophthalmic solution after cataract surgery

INTERVENTIONS:
Drug: 1. Use of preservative free diquafosol ophthalmic solution after cataract surgery — Participants are randomly assigned into the preservative free diquafosol group (Group 1), the preservative containing diquafosol group (Group 2) or the hyaluronate group (Group 3) using a simple unrestricted randomization method by the controller. The group 1 uses preservative free 3% diquafosol tetrasodium ophthalmic solution (Diquas-S; Santen Pharmaceutical Co, Ltd, Osaka, Japan) 6 times a day, the group 2 uses 3% diquafosol tetrasodium ophthalmic solution (Diquas; Santen Pharmaceutical Co, Ltd) 6 times a day and the group 3 uses 0.15% sodium hyaluronate ophthalmic solution (New Hyaluni 0.15%; Taejoon, Seoul, Korea) 6 times a day. All three groups instill each eye drop from postoperative day 1 to postoperative 12 weeks.
  Arms: Preservative free diquafosol group
Drug: 2. Use of preservative containing diquafosol ophthalmic solution after cataract surgery — Participants are randomly assigned into the preservative free diquafosol group (Group 1), the preservative containing diquafosol group (Group 2) or the hyaluronate group (Group 3) using a simple unrestricted randomization method by the controller. The group 1 uses preservative free 3% diquafosol tetrasodium ophthalmic solution (Diquas-S; Santen Pharmaceutical Co, Ltd, Osaka, Japan) 6 times a day, the group 2 uses 3% diquafosol tetrasodium ophthalmic solution (Diquas; Santen Pharmaceutical Co, Ltd) 6 times a day and the group 3 uses 0.15% sodium hyaluronate ophthalmic solution (New Hyaluni 0.15%; Taejoon, Seoul, Korea) 6 times a day. All three groups instill each eye drop from postoperative day 1 to postoperative 12 weeks.
  Arms: Preservative containing diquafosol group
Drug: 3. Use of preservative free sodium hyaluronate ophthalmic solution after cataract surgery — Participants are randomly assigned into the preservative free diquafosol group (Group 1), the preservative containing diquafosol group (Group 2) or the hyaluronate group (Group 3) using a simple unrestricted randomization method by the controller. The group 1 uses preservative free 3% diquafosol tetrasodium ophthalmic solution (Diquas-S; Santen Pharmaceutical Co, Ltd, Osaka, Japan) 6 times a day, the group 2 uses 3% diquafosol tetrasodium ophthalmic solution (Diquas; Santen Pharmaceutical Co, Ltd) 6 times a day and the group 3 uses 0.15% sodium hyaluronate ophthalmic solution (New Hyaluni 0.15%; Taejoon, Seoul, Korea) 6 times a day. All three groups instill each eye drop from postoperative day 1 to postoperative 12 weeks.
  Arms: Preservative free sodium hyaluronate group

SUMMARY:
Today, cataract surgery has become one of the safest and most effective eye surgical procedures performed on many people through the development and development of surgical techniques and instruments. However, a significant number of patients who underwent cataract surgery still complain about postoperative symptoms, such as irritation, pain, dryness, burning sensation, and foreign body sensation. The reasons of dry eye (DE) development after cataract surgery include thermal and light toxicity from the microscope, corneal epithelial damage, and frequent irrigation of ocular surface during operation, sterilization of conjunctival sac and eyelid with chemicals, transection of the corneal nerves by corneal incision, use of topical anesthetics, and preservatives in topical eye drops. In this era of high expectation of patients and premium intraocular lenses, the postoperative discomforts cannot be accepted to many patients. Several studies have recently reported that the common cause of postoperative symptoms of the patients is DE. Furthermore, if the ocular surface is deformed due to DE syndrome after surgery, the optical quality is greatly affected which results in a decrease of the quality of vision. If the tear film becomes irregular, the higher-order aberration can change due to local irregular total radius of curvature of ocular surface and result in decreased visual acuity.

There have been many attempts to treat DE syndrome after cataract surgery. Artificial tears are commonly used for the first line treatment of postoperative DE and several studies revealed its effectiveness on management of DE symptoms and signs. The postoperative use of cyclosporine 0.05 % topical eye drop improved DE symptoms and visual quality after cataract surgery. Recently, diquafosol sodium ophthalmic solution has been used for the management of DE after cataract. Diquafosol is a dinucleotide derivative and functions as agonist to the purinergic P2Y2 receptor. Diquafosol is known to stimulate not only the mucin secretion from the goblet cells but also water secretion from conjunctival epithelial cells and accessory lacrimal glands. According to previous studies, diquafosol has been found to be very effective in treating DE after cataract and to alleviate symptoms of DE syndrome. Furthermore, several studies have shown that topical diquafosol has a better efficacy in managing DE after cataract surgery than artificial tears. The preservative free diquafosol ophthalmic solution has been released recently. The use of eye drops without preservatives has also been shown to play an important role in the treatment of DE after cataract surgery. Until now, there is no study that evaluated the effect of preservative free diquafosol ophthalmic solution. Thus the investigators try to investigate the efficacy of preservative free diquafosol ophthalmic solution compared to preservative containing diquafosol ophthalmic solution and sodium hyaluronate ophthalmic solution, which are widely used in patients with DE after cataract surgery.

DETAILED DESCRIPTION:
Enrollment period : 24 months after IRB approval Participants : The subjects over 20 years old, who visited Severance hospital for cataract surgery and has dry eye. The participants who satisfies criteria, and who can be monitored at all times during each period of observation after surgery are included in the study.

Methods: The subjects are randomly divided into three groups. Group 1 will use preservative diquafosol ophthalmic solution, Group 2 will use preservative containing diquafosol ophthalmic solution, and Group 3 will use preservative free sodium hyaluronate after cataract surgery. Before surgery, all patients underwent a detailed ophthalmological examination that included evaluation of logarithm of the minimum angle of resolution (logMAR) uncorrected-distance visual acuity (UDVA) and CDVA, manifest refraction, slit-lamp examination (Haag-Streit, Köniz, Switzerland), and dry eye parameters including tear breakup time, schirmer test, OSDI, and MGD staging. All examinations were repeated at 1, and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cataract
2. age of 20 years or older
3. dry eye patient

Exclusion Criteria:

1. previous use of eye drops, except artificial tears within 3 months before cataract surgery,
2. presence of severe ocular surface diseases,
3. corneal epithelial pathologies except DE syndrome
4. a history of previous ocular surgery or trauma,

4. presence of ocular comorbidities such as glaucoma, uveitis, cystoid macular edema, 5. any surgical complications including rupture of the posterior capsule during cataract surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
1. Tear break up time (TBUT) at postoperative 3 months among the three groups. | postoperative 3 months
  1. Tear break up time (TBUT) is examined using slit lamp examination, The unit of this is "sec".
  Tear break up time (TBUT) at postoperative 3 months will be compared among the three groups.
2. Tear break up time (TBUT) changes between baseline and postoperative 3 months among the three groups. | postoperative 3 months
  2. TBUT change from baseline to postoperative 3 months will be compared among the three groups.
3. Ocular Surface Disease Index (OSDI) at postoperative 3 months among the three groups. | postoperative 3 months
  3. Ocular Surface Disease Index (OSDI) is examined using questionnaire evaluating dry eye symptom of patient (from 0 to 100). Ocular Surface Disease Index (OSDI) at postoperative 3 months will be compared among the three groups.
4. Ocular Surface Disease Index (OSDI) changes between baseline and postoperative 3 months among the three groups. | postoperative 3 months
  4. OSDI change from baseline to postoperative 3 months will be compared among the three groups.
5. Meibomian gland dysfunction (MGD) stage at postoperative 3 months among the three groups. | postoperative 3 months
  5. MGD stage is evaluated by examiner (from 0 to 4). OSDI and MGD stage is unitless. MGD stage at postoperative 3 months will be compared among the three groups.
6. Meibomian gland dysfunction (MGD) stage changes between baseline and postoperative 3 months among the three groups. | postoperative 3 months
  6 MGD stage change from baseline to postoperative 3 months will be compared among the three groups.

SECONDARY OUTCOMES:
1. The value of total higher order aberration at postoperative 3 months among the three groups. | postoperative 3 months
  1. The value of total higher order aberration is examined using iTrace aberrometer (Tracey Technologies Corp. Houston, TX). The unit of those is "μm". The value of total higher order aberration at postoperative 3 months will be compared among the three groups.
2. The change of the value of total higher order aberration between baseline and postoperative 3 months among the three groups. | postoperative 3 months
  2. The change of the value of total higher order aberration from baseline to postoperative 3 months will be compared among the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Yonsei Univeristy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baek J, Doh SH, Chung SK. The Effect of Topical Diquafosol Tetrasodium 3% on Dry Eye After Cataract Surgery. Curr Eye Res. 2016 Oct;41(10):1281-1285. doi: 10.3109/02713683.2015.1122813. Epub 2016 Apr 6. PMID 27049809
- [Background] Lee JH, Song IS, Kim KL, Yoon SY. Effectiveness and Optical Quality of Topical 3.0% Diquafosol versus 0.05% Cyclosporine A in Dry Eye Patients following Cataract Surgery. J Ophthalmol. 2016;2016:8150757. doi: 10.1155/2016/8150757. Epub 2016 Feb 16. PMID 26989503
- [Background] Park DH, Chung JK, Seo DR, Lee SJ. Clinical Effects and Safety of 3% Diquafosol Ophthalmic Solution for Patients With Dry Eye After Cataract Surgery: A Randomized Controlled Trial. Am J Ophthalmol. 2016 Mar;163:122-131.e2. doi: 10.1016/j.ajo.2015.12.002. Epub 2015 Dec 11. PMID 26685791
- [Background] Cui L, Li Y, Lee HS, Yang JM, Choi W, Yoon KC. Effect of diquafosol tetrasodium 3% on the conjunctival surface and clinical findings after cataract surgery in patients with dry eye. Int Ophthalmol. 2018 Oct;38(5):2021-2030. doi: 10.1007/s10792-017-0693-1. Epub 2017 Aug 18. PMID 28822028
- [Background] Inoue Y, Ochi S. Effects of 3% diquafosol sodium ophthalmic solution on higher-order aberrations in patients diagnosed with dry eye after cataract surgery. Clin Ophthalmol. 2016 Dec 23;11:87-93. doi: 10.2147/OPTH.S122542. eCollection 2017. PMID 28096651
- [Background] Lee H, Kim SM, Choi S, Seo KY, Kim EK, Kim TI. Effect of diquafosol three per cent ophthalmic solution on tear film and corneal aberrations after cataract surgery. Clin Exp Optom. 2017 Nov;100(6):590-594. doi: 10.1111/cxo.12521. Epub 2017 Feb 21. PMID 28222481